CLINICAL TRIAL: NCT07077577
Title: Exploring Mothers' Lived Experiences of a Holistic Birth Strategy Intervention for Labor Pain Management: A Phenomenological Qualitative Study in Southern Punjab Pakistan
Brief Title: Holistic Birth Experiences: A Qualitative Exploration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Dr. Javeria Saleem, Professor of Public Health, University of the Punjab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Holistic Approach NM
Record Dates: First submitted 2025-06-18; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Labor Pain and to Reduce Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of Holistic Approach techniques during delivery, single arm quasi experimental study (Experimental): this is single arm quasi experimental study in which intervention is given to women at time of delivery
  Interventions: Procedure: Holistic Birth Approach

INTERVENTIONS:
Procedure: Holistic Birth Approach — Holistic Birth Approach involves use of non pharmacological techniques for better labor process management with less experience of pain, fear and maternal satisfaction to women delivering the baby through normal delivery method.

SUMMARY:
This quasi experimental qualitative study aims to investigate whether Holistic Birth Approaches is useful technique for improved women's child birth experience. The study objectives include investigating the effect of holistic birth strategies on birth process and how it addresses the fear and anxiety issues during child birth. Moreover, measuring level of satisfaction among women who received holistic strategies during birth was also included in this study. Investigator will also examine the importance of holistic approach for labor pain and delivery management. The study will be conducted in chosen public healthcare facilities that either offers or gives holistic birth methods. The women in labor pain who arrived at hospital where holistic approach is offered for delivery will be included for study.

DETAILED DESCRIPTION:
The study exploration involves primarily determining the usefulness of Holistic Birth Approaches on women birth experiences especially related to labor pain, fear and anxiety challenges during child birth. Measuring Women's level of Satisfaction associates with using Holistic Birth Approaches is also another primary study objective. Further, evaluating about the factors that act as facilitators and barriers in Holistic Birth Approach implementation in Pakistan. Pregnant Women in labor pain who arrived in chosen public healthcare facilities that offers Holistic Birth Approaches for delivery will be screened for eligibility. Women willing to participate will be selected for interventional study. The included healthcare facilities must use non-clinical birth support practices such as breathing techniques, massage, hydrotherapy, aromatherapy, attendance of a midwife or doula, and emotional support for labor management.

The intervention method includes pre and post interviews. During pre-intervention interviews will be conducted to understand the women previous experiences for labor management if applicable, perceptions, knowledge about holistic approach and attitudes with respect to delivery management. Then with consent of women the holistic method will be employed during delivery for labor management. Then, after delivery post intervention interviews will be conducted to know the perceived benefits of holistic methods for women during delivery along with their intentions for future to implement or improve holistic techniques for better birth process management

ELIGIBILITY:
Inclusion Criteria:

* Pregnant reproductive age women (18-40 years) who will be willing to participate and understand Urdu language will be include in study who arrived at public health care facility for delivery and is experiencing labor pain The women from those healthcare facilities will be include that provides holistic birth approaches to women for improved birth experience particularly for labor pain, fear of birth and mother's satisfaction

Exclusion Criteria:

* Those who are not willing for interview will not be included in study. Women having serious medical condition requiring inpatient and outpatient care. Women younger than 18 and more than 40 years.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 14 (Actual)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Benefits of Holistic Birth Approach Use | Pre Intervention interviews: Pre-delivery (when women got admitted to hospital for delivery) Intervention: At time of delivery Post Intervention interviews: Post-delivery (within one or two days after delivery when women was comfortable for interviews)
  Pre Intervention; Evaluating pregnant women perspectives, experiences, knowledge and expectations before receiving any holistic birth approach Intervention Phase: Holistic Birth Approaches employed to women Post Intervention; Birth Experiences after receiving Holistic Birth Approach use

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nadia Maryam, Mphil PH, Principal Investigator — University of the Punjab
Locations (1):
- hospital from Southern Punjab, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
due to the issues of confidentiality and privacy of patients data will not be shared